CLINICAL TRIAL: NCT00345020
Title: Deep Lamellar Endothelial Keratoplasty: Small Incision Technique
Status: Withdrawn | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Vinod Mootha, MD, UTSW Medical Center at Dallas
Other Study IDs: 032005-027
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Corneal Transplantation
Keywords: Deep Lamellar Endotheliam Keratoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Deep Lamellar Endothelial Keratoplasty: Small Incision Technique

SUMMARY:
The research objectives of this study are to determine if small incision Deep Lamellar Endothelial Keratoplasty (DLEK) is able to further reduce the degree of corneal astigmatism and shorten the time course of corneal topography stabilization compared to standard full thickness corneal transplant (PKP) surgery.

DETAILED DESCRIPTION:
Split thickness lamellar corneal transplants have been performed for many years to replace the front part of the cornea and have been highly successful. What is different about this study is that the surgical procedure involves replacement of the back layers of the cornea rather than the front layers of the cornea. This replacement is done through a small pocket incision to avoid changes in the front surface of the cornea. By leaving the front surface in the cornea without sutures or incisions there is felt to be an advantage in healing and recovery time for the patient. In addition, this particular study will use a pocket incision that is even shorter and smaller in length than the one used in previous DLEK surgeries to try to make healing time even faster and more predictable. This procedure has been successfully performed on patients in the Netherlands for over five years. The procedure has also been successfully performed by doctors in the United States. Subjects participating in this study will be among the first patients to undergo this procedure in the The University of Texas Southwestern Medical Center at Dallas.

ELIGIBILITY:
Inclusion Criteria: Subjects enrolled in this study will have endothelial dysfunction to a level generally accepted as requiring standard PKP for treatment. Subjects will be offered the alternative surgery of this protocol. All subjects will be between the ages of 21 and 95. Males and females are eligible.

-

Exclusion Criteria: Central corneal scars, presence of a filtering bleb and uncontrolled glaucoma.

-

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
to determine if small incision Deep Lamellar Endothelial Keratoplasty (DLEK) is able to further reduce the degree of corneal astigmatism and shorten the time course of corneal topography stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Mootha, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States